CLINICAL TRIAL: NCT05936619
Title: MindEx: A Novel, Multifocal, Cognitive Brain-Machine Interface System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nader Pouratian (Other)
Responsible Party: Sponsor-Investigator, Nader Pouratian, Professor & Chair, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU-2023-0306
Record Dates: First submitted 2023-05-25; First posted 2023-07-10 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Paralysis; Quadriplegic
Keywords: spinal cord injury; brain-computer interface; brain-machine interface
MeSH Terms: conditions — Paralysis; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Mind Extender (MindEx) (Experimental): MindEx consists of two Neuroport Multi-Port Arrays, described in detail in the intervention description. Each NeuroPort Multi-Port Array comprises two electrode arrays implanted into human brain tissue, for a total of four electrode arrays. These will be in 1) prefrontal cortex, a brain area involved in scene comprehension, action selection, and error signaling, 2) premotor cortex, a brain area involved in planning ongoing and upcoming actions, 3) posterior parietal cortex, a brain area involved in processing sensory-to-motor transformations during movements, and 4) primary motor cortex, responsible for controlling movement. The pair of electrode arrays in each NeuroPort Multi-Port Array connect to a single percutaneous pedestal attached to the skull during a surgical procedure. Following recovery from the surgical placement, subjects will participate in study sessions up to 5 times a week. They will learn to use thought to control applications on a computer, a laptop, or a tablet.
  Interventions: Device: Mind Extender (MindEx)

INTERVENTIONS:
Device: Mind Extender (MindEx) — NeuroPort Multi-Port Arrays allow for the local recording of cerebral cortex. The Mind Extender (MindEx) system is primarily composed of two NeuroPort Multi-Port Arrays. Each Multi-Port device consists of two arrays, each with 100 electrodes in a 10 x 10 configuration, with dimensions 4 mm x 4 mm x 1.5 mm (W x H x D), and a titanium percutaneous connector, 19 mm diameter at the base. Each MultiPort can have a total of 128 active channels (capable of transmitting neural signals to the percutaneous connector) across the two arrays. In our design, we will split active channels evenly between the two arrays resulting in 64 active channels per array. The four arrays of the two Multi-Port device will be implanted into prefrontal cortex, premotor cortex, primary motor cortex, and posterior parietal cortex.

SUMMARY:
This research study is being done to develop a novel brain-computer interface (BCI) technology that can enable severely paralyzed individuals to interact with the world through direct brain-control of a computer. This technology is named MindEx (for Mind Extender). It utilizes four implanted "chips" in the human brain from which investigators can record brain activity during subjects' thoughts and decode meaningful information from this activity to be used as control signals for a computer, a laptop, or a tablet. The use of four brain regions is a significant differentiating feature and scientific innovation of this study over much prior work in this space, that typically derived control signals from one, or sometimes two brain regions. The brain regions to be used here can allow the decode of multiple variables simultaneously, including not just moment-to-moment position, but also high-level goals, intentions, decisions, scene comprehension, and error-related signals involved in natural human behavior. The research is being done through a prospective, longitudinal, single-arm early feasibility study to examine the safety and effectiveness of using MindEx to provide the user an intuitive, efficient, and accurate ability to control multiple applications on a computer interface such as a word processor, a paint application, or to play simple video games. Such versatility could greatly improve the autonomy and quality of life of severely paralyzed individuals. Two subjects will be enrolled, each implanted with MindEx for a period of at least 53 weeks and up to 313 weeks. The study is expected to take at least one year and up to six years in total.

ELIGIBILITY:
Inclusion Criteria:

* Paralysis resulting from cervical spinal cord injury (SCI), brainstem stroke (ischemic or hemorrhagic), or amyotrophic lateral sclerosis (ALS)
* Provide informed consent
* Understand and comply with instructions, if necessary, with the aid of a translator
* Communicate via speech or other means
* Surgical clearance
* Life expectancy greater than 12 months
* Travel to study locations up to five days per week for the duration of the study
* Caregiver monitor for surgical site complications and behavioral changes on a daily basis
* Psychosocial support system
* Stable ventilator status

Exclusion Criteria:

* Presence of memory problems
* Intellectual impairment
* Psychotic illness or chronic psychiatric disorder, including major depression if untreated
* Poor visual acuity
* Pregnancy
* Active infection or unexplained fever
* Scalp lesions or skin breakdown
* HIV or AIDS infection
* Active cancer or chemotherapy
* Diabetes
* Autonomic dysreflexia
* History of seizure
* Implanted hydrocephalus shunt
* Prior cranioplasty
* Other implanted devices
* Medical conditions contraindicating surgery and chronic implantation of a medical device
* Unable to undergo MRI or anticipated need for MRI during the study
* Breastfeeding an infant (direct nursing or via a bottle of expressed milk)
* Chronic oral or intravenous use of steroids or immunosuppressive therapy
* Suicidal ideation
* Drug or alcohol dependence
* Planning to become pregnant, or unwilling to use adequate birth control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Continuous trajectory decoding | Six years after array implantation
  A primary objective of this study is to evaluate the effectiveness of the system in providing users the ability to continuously move a cursor on a tablet/computer.
  The hypothesis is that trajectory readability from neural signals will be significantly greater than the level of chance.
  Standardized tests will be used to test this objective, and performance will be compared to the level of chance.
  One example of a standardized test to be used is the accuracy of continuous trajectory decoding measured by the radial-8 assessment task.
Incidence of intervention-related adverse events | Six years after array implantation
  Serious adverse events (SAE) will be evaluated against a 1% threshold level. We will use regular inspection of the subjects' scalps to assess for breakdown, discharge, or infection, and use history and physical exam to evaluate for new symptoms, and compare to baseline assessments.
Competency in computer/tablet control | Six years after array implantation
  An underlying hypothesis in this study is that the system will enable users the ability to control a computer/tablet interface by selecting icons.
  An underlying hypothesis in the study is that neural signals will enable decoding the chosen target at higher accuracy than the level of chance.
  Standardized tests will be used to test this objective, and performance will be compared to the level of chance.
  An example of a standardized test to be used is the brain-control for tablet test (BCTT) which grades the accuracy of target selection by mental fixation to the level of chance.
Efficacy of multiple brain regions for neural control over subsets of brain regions | Six years after array implantation
  An objective of this study is to determine whether the combination of neural signals from multiple brain regions in brain-computer interface control is more advantageous than from a subset of the brain regions being tested.
  The hypothesis is that because the four brain regions being implanted each encode different cognitive functions, their integration will be more useful to brain-computer interface control, than any subset of these regions.
  This objective will be tested by standardized tests (such as those mentioned for "Competency in computer/tablet control" and "Continuous trajectory decoding") in different groups of brain regions and reported for each, such as:
  1. All four brain regions: prefrontal cortex (PFC), posterior parietal cortex (PPC), dorsal premotor cortex (PMd), primary motor cortex (M1)
  2. PMd,PPC, and M1
  3. PPC and M1 alone

SECONDARY OUTCOMES:
Change in quality of life | Time Frame: Annually, for six years
  The functional change in quality of life will be evaluated through a Quality-of-Life Inventory (QOLI) administered periodically throughout the study. This is a 32-item questionnaire with a score range from 1-77, with higher scores reflecting higher satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Investigators with established research programs will be eligible for data sharing. Interested investigators will be required to submit a summary of the proposed work and requested data elements. If approved by the Principal Investigator of the study, data will be shared. This data will be de-identified and coded. There is no plan to share identifiers outside the study team.